CLINICAL TRIAL: NCT06994572
Title: A Phase 1, Open-Label, Dose Escalation, and Dose Expansion Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CT-01 as Monotherapy and Combination Therapy With Everolimus in Subjects With Intermediate or Advanced Hepatocellular Carcinoma (BCLC Stage B or C) With Preserved Liver Function (Child-Pugh Class A)
Brief Title: Study of CT-01 as Monotherapy and Combination Therapy in Subjects With Intermediate or Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Captor Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT-01-CD-1
Record Dates: First submitted 2025-04-29; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CT-01 PART 1A: Monotherapy - Dose Escalation (Experimental): Subjects receive CT-01 monotherapy at predefined dose levels. Doses assigned according to a dose-escalation protocol.
  Interventions: Drug: CT-01
- CT-01 PART 1B: Monotherapy - Dose Expansion (Experimental): Subjects receive CT-01 monotherapy at the selected recommended dose level identified in Part 1A
  Interventions: Drug: CT-01
- CT-01 PART 2A: Combotherapy - Dose Escalation (Experimental): Subjects receive CT-01 and everolimus orally once daily in 28-day cycles
  Interventions: Drug: CT-01; Drug: EVEROLIMUS
- CT-01 PART 2B: Combotherapy - Dose Expansion (Experimental): Subjects receive CT-01 and everolimus at the recommended combination dose.
  Interventions: Drug: CT-01; Drug: EVEROLIMUS

INTERVENTIONS:
Drug: CT-01 — Investigational small-molecule degrader targeting transcription factors in HCC. Used as monotherapy or with everolimus in dose-escalation/expansion settings. Specific to protocol CT-01-CD-1.
Drug: EVEROLIMUS — Approved mTOR inhibitor used in combination with CT-01 for HCC in this study. Evaluated for safety, tolerability, and PK/PD in CT-01-CD-1 protocol.
  Arms: CT-01 PART 2A: Combotherapy - Dose Escalation; CT-01 PART 2B: Combotherapy - Dose Expansion

SUMMARY:
This is a Phase 1, open-label, multicenter, dose-escalation and dose-expansion study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of CT-01, administered either as monotherapy or in combination with everolimus. The study population includes subjects with intermediate or advanced hepatocellular carcinoma (HCC) who have progressed on, or are intolerant to, at least one prior line of systemic treatment. All available standard-of-care therapies should have been received, if deemed appropriate by the investigator (unless contraindicated or considered inappropriate by the treating physician). Eligible subjects are classified as Barcelona Clinic Liver Cancer (BCLC) stage B or C and must not be amenable to curative treatment approaches. Only subjects with preserved liver function (Child-Pugh Class A, score 5-6) at screening are eligible. Approximately 141 participants will be enrolled across 20 sites in Europe (France, Spain, and Germany).

DETAILED DESCRIPTION:
This is an open-label, multicenter study evaluating the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of CT-01 in subjects with advanced hepatocellular carcinoma (HCC). The study consists of two sequential parts.

Part 1 investigates CT-01 as monotherapy and includes a dose-escalation phase (Part 1A) followed by a dose-expansion phase (Part 1B). A Bayesian Optimal Interval (BOIN) design will be used, with up to seven predefined dose levels. Additional subjects may be enrolled to backfill dose levels of interest. Treatment will be administered in 28-day cycles, with dose-limiting toxicities (DLTs) assessed during Cycle 1. Dose decisions will be made by an Independent Data Monitoring Committee (IDMC), with input from a Safety Monitoring Committee (SMC).

Part 2 evaluates CT-01 in combination with everolimus and includes a dose-escalation phase (Part 2A) and a dose-expansion phase (Part 2B). Up to four dose levels are planned in Part 2A, with starting doses informed by Part 1 results. As in Part 1, DLTs will be assessed during Cycle 1 and reviewed by the IDMC and SMC.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to provide informed consent and able to comply with the study procedures and restrictions.
* Are ≥18 years of age and of any gender at the time of screening.
* Have confirmed histological and/or radiological diagnosis of HCC with a Child-Pugh Class A score of 5 to 6 points within 7 days of first dose of study drug.
* Has BCLC stage B and are ineligible for or are refractory to locoregional therapy and not amenable to a curative treatment approach, or BCLC stage C and are not amenable to a curative treatment approach.
* Have progressed on or are intolerant to ≥1 prior systemic standard of care treatment. All available standard of care treatments should have been received as prior systemic treatment if deemed appropriate by the investigator (unless such treatments are deemed contraindicated or inappropriate by the treating physician).
* Have Eastern Cooperative Oncology Group (ECOG) score ≤1.
* Have at least one measurable disease lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and/or modified RECIST (mRECIST), with a minimum of 1 target lesion in the liver at screening.
* Female subjects may be enrolled if they refrain from donating eggs (ova, oocytes) for the purpose of reproduction during the treatment period and for 6 months after the treatment period and if they are:

  1. Documented to be surgically sterile or postmenopausal, or
  2. Practicing true abstinence for at least 28 days prior to investigational medical product (IMP) administration and for 6 months after the treatment period and having a negative pregnancy test prior dosing, or
  3. Willing and able to comply with two forms of contraception methods, including one physical barrier (condom or diaphragm) plus another method, such as adequate hormonal method (eg, contraceptive implants, injectables, oral contraceptives) or nonhormonal methods (eg, intrauterine device, spermicidal) during and for 6 months after the treatment period and having a negative pregnancy test prior dosing. Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male subjects with female partners of childbearing potential may be enrolled if they refrain from donating sperm during the treatment period and for 6 months after the last IMP administration and if they are:

  1. Documented to be surgically sterile (vasectomy), or
  2. Practicing true abstinence during the treatment period and for 6 months after the last IMP administration, or
  3. Willing and able to comply with two forms of contraception methods, including one physical barrier (condom or diaphragm) during the treatment period and for 6 months after the last IMP administration. Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Have not recovered from toxicities to baseline or Grade ≤1 by CTCAE version 5.0 from prior anticancer therapy, except alopecia and sub-optimally treated nausea, vomiting, or diarrhea.
* Have a history of liver transplant.
* Any other active malignancy at time of screening or diagnosis of another malignancy within 2 years before screening that requires active treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.
* Have central nervous system (CNS) metastases or any other Grade >2 CNS disorder. Subjects with CNS metastases who are stable on their treatment since a minimum of 4 weeks prior to screening are eligible.
* Have recent esophageal or gastric variceal bleeding within 4 weeks prior to screening. Subjects with treated, stable, or small varices without bleeding within the 4 weeks prior to screening are eligible.
* Have a history of symptomatic ascites requiring paracentesis within the past 3 months prior to screening.
* Have a prior diagnosis of rhabdomyolysis from any cause.
* Subjects with known retinal disease (eg, diabetic retinopathy, macular degeneration, retinal detachment/tear, etc).
* Have a history of clinically significant cytokine release syndrome as assessed by the treating physician, clinically significant hypotension (defined as a blood pressure [BP] consistently <90/60 mmHg and/or a BP associated with symptoms of hypotension (dizziness, fainting, orthostatic hypotension [systolic BP drop of >20 mmHg or diastolic BP drop of >10 mmHg on orthostasis]), symptomatic hypocalcemia and/or a calcium level <1.5 mmol/L.
* Have a history of pneumonitis or pericarditis.
* Subjects who are not, in the opinion of the investigator, willing or able to comply with the protocol or who present a contraindication to any study procedure.
* Have inadequate hematologic and end-organ function, defined as follows:

  * Hemoglobin <8.5 g/dL
  * Absolute neutrophil count <1,500 per mm3
  * Platelet count <75,000 per mm3
  * Total bilirubin >2 × ULN for the designated testing laboratory
  * AST or ALT >5 × ULN
  * Serum creatinine >1.5 × ULN
  * International normalized ratio (INR) >1.7 × ULN
  * Glomerular filtration rate (GFR) < 50 mL/min
* Have imaging findings corresponding to HCC with ≥50% liver occupation, or clear invasion into the bile duct.
* Have an active infection with the hepatitis B virus (HBV) or hepatitis C virus (HCV).

  1. Patients with acute hepatitis B infection are excluded. Acute Hepatitis B is defined based on the following serology profile: positive hepatitis B surface antigen (HBsAg positive), positive total hepatitis B core antibody (anti-HBc positive), IgM antibody positive to hepatitis B core antigen (IgM anti-HBc positive), and hepatitis B surface antibody negative (anti-HBs negative) test at screening.
  2. Patients with a past or resolved HBV infection (defined as HBsAg positive and anti-HBc positive) are eligible.
  3. Patients positive for HCV antibody are eligible only if PCR is negative for HCV ribonucleic acid (RNA).
  4. Chronic HBV (HBsAg positive, undetectable or low HBV DNA, and normal ALT) is eligible if patients are receiving direct-acting antiviral treatment.
  5. Patients with resolved hepatitis C infection are eligible. This is defined as undetectable or unquantifiable HCV RNA 12 weeks or longer after treatment completion (defined as a sustained virological response).
  6. Patients with untreated HCV infection or have not completed treatment for HCV infection.
  7. Patients with treated HCV infection but with a HCV viral load above the level of quantification.
* Have a history of human immunodeficiency virus (HIV) infection.
* Have life expectancy shorter than 3 months.
* Have received any systemic anticancer treatment or any investigational treatment within 14 days or at least 5 half-lives of the treatment, whichever is shorter, prior to screening.
* Are unable to take oral medications.
* Have a known malabsorption syndrome.
* Applicable to subjects enrolling in Part 2 only:

  * Are currently receiving treatment with the cytochrome P450 (CYP) 3A4 inhibitors (eg, azoles, clarithromycin, or grapefruit), CYP3A4 inducers (eg, rifampin, carbamazepine, phenytoin, or St. John's wort), or p-glycoprotein (P-gp) inhibitors or inducers (eg, verapamil, quinidine, amiodarone, diltiazem, erythromycin, cyclosporine, ketoconazole, ritonavir, or tamoxifen).

Subjects able to receive modified dose of the P-gp or CYP3A4 inhibitors based on everolimus drug label may be eligible at the discretion of the investigator in consultation with the sponsor and Medical Monitor.

* Have a known intolerance or hypersensitivity to everolimus, its component (eg, lactose), or other rapamycin derivatives.
* Subjects who are planned for elective surgery within 56 days of planned treatment Day 1 are excluded due to the risk of impaired wound healing with everolimus and the requirement to interrupt everolimus treatment per the everolimus SmPC. (Note: subjects who can delay elective surgery beyond Day 56 (Week 8, RECIST version 1.1 assessment) of study treatment are eligible for the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2029-04-16 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) during CT-01 monotherapy | Up to 12 months
  Safety and tolerability of CT-01 will be evaluated by monitoring the incidence of TEAEs, SAEs, AESIs, and TEAEs leading to study discontinuation or death.
  Unit of Measure: Number, nature, sverity and relation plausibility of AE
Maximum tolerated dose (MTDm) of CT-01 monotherapy | Up to 12 months
  The MTDm will be determined based on the incidence and type of dose-limiting toxicities (DLTs) during Cycle 1 of CT-01 monotherapy.
  Unit of Measure: mg/day
Number of participants with treatment-emergent adverse events (TEAEs) during CT-01 and everolimus combination therapy | Up to 12 months
  Safety and tolerability will be assessed through monitoring of TEAEs, SAEs, AESIs, and TEAEs leading to study discontinuation or death during combination therapy.
  Unit of Measure: Number, nature, sverity and relation plausibility of A
Maximum tolerated dose (MTDc) of CT-01 in combination with everolimus | Up to 12 months
  The MTDc will be determined based on the incidence of DLTs during Cycle 1 of the combination therapy.
  Unit of Measure: mg/day

SECONDARY OUTCOMES:
Objective response rate (ORR) per RECIST v1.1 and mRECIST for CT-01 monotherapy | Up to 12 months
  Proportion of participants achieving complete or partial response as per RECIST v1.1 and mRECIST.
  Unit of Measure: Percentage of participants
Objective response rate (ORR) per RECIST v1.1 and mRECIST for CT-01 and everolimus | Up to 12 months
  Proportion of participants achieving complete or partial response during combination therapy.
  Unit of Measure: Percentage of participants
Maximum plasma concentration (Cmax) | Up to 12 months
  Cmax will be determined for CT-01 using non-compartmental analysis. Unit of Measure: ng/mL
Area under the concentration-time curve (AUC) | Up to 12 months
  AUC will be calculated for active metabolite of CT-01 using non-compartmental methods (AUC₀-t and AUC₀-inf).
  Unit of Measure: ng·h/mL
Time to maximum concentration (Tmax) | Up to 12 months
  Tmax will be recorded as the time to reach Cmax for CT-01. Unit of Measure: Hours
Change from baseline in MELD-Na score during combination therapy | Up to 12 months
  Change in MELD-Na score (range: typically 6 to 40; higher scores indicate worse liver function) from baseline during CT-01 and everolimus treatment. Unit of Measure: score
Change from baseline in Child-Pugh score during combination therapy | Up to 12 months
  Change in Child-Pugh score (range: 5-15; higher scores indicate worse liver function) from baseline during CT-01 and everolimus treatment.
  Unit of Measure: score
Change from baseline in Albumin-Bilirubin (ALBI) score during combination therapy | Up to 12 months
  Change from baseline in ALBI score will be evaluated during CT-01 and everolimus combination therapy. The ALBI score is calculated using serum bilirubin and albumin. Changes from baseline will be summarized by time point. Higher scores indicate worse liver function.
  Unit of Measure: score
Change from baseline in lipid profile during combination therapy | Up to 12 months
  Change in serum lipid parameters (total cholesterol, LDL, HDL, triglycerides) from baseline during CT-01 and everolimus treatment.
  Unit of measure: mmol/L
Change from baseline in serum glucose levels during combination therapy | Up to 12 months
  Change in blood glucose concentration from baseline during CT-01 and everolimus treatment.
  Unit of Measure: mmol/L
Change from baseline in serum alpha-fetoprotein (AFP) levels during combination therapy | Up to 12 months
  Change in serum AFP concentration from baseline during treatment with CT-01 in combination with everolimus. AFP is a tumor marker used in hepatocellular carcinoma.
  Unit of Measure: ng/mL
Terminal half-life (T1/2) | Up to 12 months
  T1/2 will be estimated for active metabolite of CT-01 from the log-linear terminal phase of the concentration-time curve.
  Unit of Measure: Hours
Title: Maximum plasma concentration (Cmax) | Up to 12 months
  Cmax will be determined for CT-01 in combination with everolimus using non-compartmental analysis.
  Unit of Measure: ng/mL
Change from baseline in serum glucose levels during monotherapy | Up to 12 months
  Change in blood glucose concentration from baseline during CT-01 monotherapy. Unit of Measure: mmol/L
Area under the concentration-time curve (AUC) | Up to 12 months
  AUC for active metabolite of CT-01 in combination with everolimus will be calculated using non-compartmental methods.
  ng·h/mL
Time to maximum concentration (Tmax) | Up to 12 months
  Tmax will be recorded for CT-01 when administered with everolimus. Unit of Measure: Hours
Terminal half-life (T1/2) | Up to 12 months
  T1/2 will be estimated for active metabolite of CT-01 in combination therapy using non-compartmental analysis.
  Unit of Measure: Hours
Change from baseline in lipid profile during monotherapy | Up to 12 months
  Change in serum lipid parameters (total cholesterol, LDL, HDL, triglycerides) from baseline during CT-01 monotherapy.
  Unit of Measure: mmol/L
Change from baseline in Albumin-Bilirubin (ALBI) score during monotherapy | Up to 12 months
  Change from baseline in ALBI score will be evaluated during CT-01 monotherapy. The ALBI score is calculated using serum bilirubin and albumin. Changes from baseline will be summarized by time point. Higher scores indicate worse liver function.
  Unit of Measure: score
Change from baseline in Child-Pugh score during monotherapy | Up to 12 months
  Change in Child-Pugh score (range: 5-15; higher scores indicate worse liver function) from baseline during CT-01 monotherapy.
  Unit of Measure: score
Change from baseline in MELD-Na score during monotherapy | Up to 12 months
  Change in MELD-Na score (range: typically 6 to 40; higher scores indicate worse liver function) from baseline during CT-01 monotherapy.
  Unit of Measure: score
Change from baseline in serum alpha-fetoprotein (AFP) levels during monotherapy | Up to 12 months
  Change in serum AFP concentration from baseline during CT-01 monotherapy. AFP is a tumor marker used in hepatocellular carcinoma.
  Unit of Measure: ng/mL

OTHER OUTCOMES:
Changes in ISR gene expression (ATF3, DDIT3) during CT-01 monotherapy | Up to 12 months
  mRNA expression levels measured by qPCR as pharmacodynamic markers. Unit of Measure: Relative mRNA expression (ΔCt or fold change)
Association between PK/PD and anti-tumor activity during CT-01 monotherapy | Up to 12 months
  Correlation analysis between drug exposure (PK) and PD biomarkers with objective tumor response.
  Unit of Measure: Correlation coefficient (r)
Changes in GSPT1 and NEK7 protein levels during CT-01 and everolimus combination therapy | Up to 12 months
  Evaluation of protein modulation in PBMCs following CT-01 and everolimus administration.
  Unit of Measure: Relative expression (fold change)
Changes in ISR gene expression (ATF3, DDIT3) during CT-01 and everolimus combination therapy | Up to 12 months
  ISR-related gene expression changes assessed via qPCR in PBMCs or blood. Unit of Measure: Relative mRNA expression (ΔCt or fold change)
Association between PK/PD and anti-tumor activity during CT-01 and everolimus combination therapy | Up to 12 months
  Analysis of correlation between PK exposure and PD effects with observed tumor response.
  Unit of Measure: Correlation coefficient (r)
Changes in GSPT1 and NEK7 protein levels during CT-01 monotherapy | Up to 12 months
  Protein levels assessed in PBMCs by western blot as indicators of target engagement.
  Unit of Measure: Relative expression (fold change)